CLINICAL TRIAL: NCT01121601
Title: Effectiveness and Tolerance of CoSeal in the Prevention of Hepatic Adherences of Novo Post Operational Within the Framework of a Hepatic Surgery of Resection in Two Times for Hepatic Metastases: Study of Phase II/III.
Brief Title: CoSeal in Liver and Biliary Surgery in Prevention of Denovo Hepatic Adhesion
Acronym: COLIBIS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Practices in surgery have evolved and the study has not interest yet
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P/2010/94
Record Dates: First submitted 2010-05-04; First posted 2010-05-12 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Patient With Hepatic Metastasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group COSEAL (Experimental)
  Interventions: Procedure: hepatic surgery of resection
- Reference group (Active Comparator)
  Interventions: Procedure: hepatic surgery of resection

INTERVENTIONS:
Procedure: hepatic surgery of resection — after metastasis liver resection , Coseal will be administered at 4 mL by dose, administration of 1 to 3 dose in fontion of liver adherence Coseal will be administered by spray at 5 to 10 cm of liver.
  Arms: Group COSEAL
Procedure: hepatic surgery of resection — this is a liver metastasis resection according to liver chirurgical guidelines study drug not administered in this group
  Arms: Reference group

SUMMARY:
Study of phase II: Clinical study national, exploratory, multicentric, prospective, randomized, as a double blind man evaluating the effectiveness and the tolerance of the treatment by a surgical gel of sealing containing polyethylene glycol in the prevention of operational adherences post.3 Study of phase III: Clinical study national, multicentric, prospective, randomized, controlled, as a double blind man comparing a group controls with a group of patients treated by a surgical gel of sealing containing polyethylene glycol in the prevention of hepatic adherences of novo post operational.

ELIGIBILITY:
Inclusion Criteria:

* Major patients.
* Hepatic Carriers of metastases.
* Eligible with a procedure of surgical eradication in two brought closer times (time lower than 3 months).
* Strategy validated in multidisciplinary meeting of cancerology.
* Enlightened Assent given and signed before the intervention.

Exclusion Criteria:

* Anaesthetic Counter-indications with a procedure in two times
* Carcinose péritonéale, reached metastatic not éradicable
* Over-sensitiveness or allergy known to polyethylene CoSeal glycol
* Concomitant Use of another antiblocking agent
* Immunodéprimés Patients or taking drugs immunodépresseurs with the long court like the corticosteroids,
* Impossibility of subjecting itself to the medical monitoring imposed by the study for reasons geographical, social, psychic or medical.
* Concomitant Participation in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-08

PRIMARY OUTCOMES:
HEPATIC ADHERENCE SEVERITY | 3 years
  Measure of hepatic adherence :
  SCORE 0: NO HEPATIC ADHERENCE SCORE 1: SHADOW ON HEPATIC ADHERENCE SCORE 2: VASCULAR OR DENSE HEPATIC ADHERENCE SCORE 3:COHESIVE HEPATIC ADHERENCE SCORE 4: DISSECTION IN ANOTHER PLAN
  THIS 5 SCORE WILL BE ANALYSED ON THE 8 SEGMENT AND ON PEDICLE OF LIVER

SECONDARY OUTCOMES:
LIVER RELEASE VALUE | 3 years
  DISSECTION PHASE BETWEEN INCISION AND PARTIAL OR TOTAL EXPOSITION OF LIVER
LOSS OF BLOOD | 3 years
CoSeal tolerance | 3 years
per operative complication | 3 years
post operative complication | 3 years
hospitalisation time | 3 years
operative difficulty | 3 years
  score 0 if there are no difficulty for the release of liver or score 10 if dissection of liver is impossible
de novo hepatic adherence extension | 3 years
  0 : no extension of hepatic adherence
  1. : 1/3 of area affected
  2. : between 1/3 and 2/3 of area affected
  3. : more than 2/3 of area affected
hepatic adherence reformation | 3 years
adherence composite score | 3 years
  this is a mathematic score in relation with area and severity of liver adherence
composite score and surgery difficulty | 3 years
  this is a correlation between the composite score, the morbidity criteria and dissection difficulty
liver adherence score validation | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruno HEYD, PU-PH, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France, France